CLINICAL TRIAL: NCT04230460
Title: Cannabis Impairment Detection Application (CIDA)
Acronym: CIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Brain Monitoring, Inc. (Industry)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: N44DA-19-1218
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Driving Under the Influence; Marijuana Intoxication; Alcohol Intoxication
Keywords: Marijuana; Cannabis; Alcohol; Driving; DUI; Drinking behavior; Substance Use; Driving Impairment; Drugs; EEG; SDLP
MeSH Terms: conditions — Driving Under the Influence; Alcoholic Intoxication; Marijuana Abuse; Drinking Behavior; Substance-Related Disorders | interventions — nabiximols; Dronabinol; Inhalation; Ethanol

STUDY DESIGN:
Intervention Model Description: The University of Iowa study is a counter-balanced dose-response protocol where all participants will receive all three doses of marijuana (plus alcohol if they qualify).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: University of Iowa: Triple (Participant, Investigator, Outcomes Assessor) blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0% THC/ 0% CBD (Placebo Comparator)
  Interventions: Drug: Cannabis (THC) (Inhaled) Placebo
- THC (5-10% [37.5 mg]) / Low CBD (<1% [2.5 mg]) (Experimental)
  Interventions: Drug: Cannabis (High% THC) (Inhaled)
- THC (>10% [62.5 mg]) / Low CBD (<1% [2.5 mg]) (Experimental)
  Interventions: Drug: Cannabis (Very High% THC) (Inhaled)
- 0.065% BAC (Experimental)
  Interventions: Drug: Alcohol (oral)

INTERVENTIONS:
Drug: Cannabis (THC) (Inhaled) Placebo — Cannabis vapor is produced from 500 mg of dried plant material (placebo) (0% THC). Participants will inhale ad libitum over 10 minutes.
  Other Names: Marihuana; Marijuana
  Arms: 0% THC/ 0% CBD
Drug: Cannabis (High% THC) (Inhaled) — Cannabis vapor is produced from 500 mg of dried plant material (7.5% THC). Participants will inhale ad libitum over 10 minutes.
  Other Names: Marihuana; Marijuana
  Arms: THC (5-10% [37.5 mg]) / Low CBD (<1% [2.5 mg])
Drug: Cannabis (Very High% THC) (Inhaled) — Cannabis vapor is produced from 500 mg of dried plant material (12.5% THC). Participants will inhale ad libitum over 10 minutes.
  Other Names: Marihuana; Marijuana
  Arms: THC (>10% [62.5 mg]) / Low CBD (<1% [2.5 mg])
Drug: Alcohol (oral) — Subjects will be dosed to achieve a 0.05% Blood Alcohol Concentration (BAC), so the amount of alcohol consumed will be calculated to produce a peak BAC of 0.065%. Subjects will be served three equal-sized drinks, 10-minutes apart, and be instructed to pace each drink evenly over the 10-minute period.
  Other Names: Ethanol; Ethyl Alcohol
  Arms: 0.065% BAC

SUMMARY:
Subjects will participate in a 4-visit study protocol in which they will be asked to complete a set of computerized tasks and a 45-minute simulated drive in a driving simulator. Subjects will be administered marijuana of varying pre-determined concentrations of delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) during 3 of the visits and alcohol during one of the visits. Throughout the duration of each visit, brain activity will be measured noninvasively using an electroencephalogram (EEG) headset.

The purpose of this study is to:

1. Further understand the effects of acute cannabis intoxication on driving performance in a driving simulator
2. Develop and refine brain-based biomarkers of impairment due to acute cannabis intoxication

DETAILED DESCRIPTION:
At the University of Iowa, subjects who currently use cannabis recreationally (> once a month but < 5 times a week) will be recruited. They will then undergo a screening visit in which consent is obtained, questionnaires are given, and a physical exam is administered. They will then be scheduled for their next 3 (or 4 if participating in the alcohol arm), which will be at least one week apart. At each visit, in counter-balanced manner, subjects will be administered 500 mg of either placebo Marijuana (trace amounts of THC), high THC marijuana (7.5%), or very high THC marijuana (12.5%). All marijuana will be inhaled ad libitum via a Volcano® Digit vaporizer. Additionally, a subset of subjects will be asked to complete a fourth study visit that administers alcohol in place of cannabis. As subjects complete the third study visit and meet criteria for the alcohol arm, they will be invited to participate in the fourth study visit until eighteen subjects complete the study's alcohol arm. After drug administration, subjects will be asked to complete a set of computerized neurocognitive tasks (1 hour), followed by a simulated drive (45 minutes).

Throughout the duration of each visit, EEG will be collected. EEG is a non-invasive method of recording the electrical activity of the brain. Additionally, blood draws will be taken at pre-determined time points.

Finally, subjects will be monitored until the drug effects have subsided sufficiently to ensure it is safe to transport them home. Subjects will be transported home.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 50 years of age in good health (21 to 50 for alcohol arm)
* Valid US driver's license and have been licensed driver for two years
* Restrictions on driver's license limited to vision correction only
* Drive at least three times per week
* Must be able to drive without special or non-standard equipment
* Must be able to attend three morning daytime study visits lasting approximately 5 to 6 hours
* Must be willing to abstain from alcohol use in the day prior to their study appointments
* Must be willing to abstain from use of their own cannabis while enrolled in the study
* Live within 1-hour driving radius of National Advanced Driving Simulator (NADS)
* Must currently use cannabis at least once every three months and no more than four times per week (must be current user)
* Peripheral veins suitable for venipuncture
* Blood pressure within clinically normal range
* If invited to complete alcohol arm: Must be considered a light or moderate drinker according to Quantity-Frequency-Variability Scale (QFV) or, if a heavy drinker, not drink more than 1-2 times a week and not have a modal quantity of 5-6 drinks

Exclusion Criteria:

* Females who are pregnant or test positive for pregnancy or are breastfeeding
* Any known sleep disorders, or family history of sleep disorders
* Any neurological or pulmonary disorders (or taking medications for such)
* Any psychiatric disorder (or taking medications for such)
* Any eating disorders
* Recent (past 5 years) head injury, or older head injury with current symptoms
* High blood pressure, Heart disease, diabetes, or history of stroke or taking medications to treat
* Any known behavioral or attention disorder (or taking medications for such)
* Untreated/Untreatable vision or auditory issues (because testing currently requires both senses)
* Excessive tobacco use (more than 10 cigarettes a day)
* Excessive caffeine use (5 or more servings per day)
* Excessive alcohol (20 or more drinks per week)
* Donation of 450 mL or more of blood in the two weeks preceding study drug administration
* Regular use of pain medications other than over-the-counter
* Any medication use that causes drowsiness or is contraindicated for driving
* Use of prescription drugs not prescribed to them or illicit drugs other than cannabis
* Propensity to motion sickness (more than 2-3 episodes where intensity is moderate or above)
* History of substance abuse or substance addiction
* Currently participating in or interested in drug abuse treatment, or participation in a program in past 60 days
* Current cannabis use disorder or alcohol use disorder [as determined by scores on the Cannabis Use Disorder Identification Test (CUDIT) and Alcohol Use Disorder Identification Test (AUDIT)]

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Driving Performance | Through entire 45-minute drive, 0.5-1.3 hour post cannabis administration
  Measured by standard deviation of lane position (SDLP, a gold standard metric of driving performance, O'Hanlon, 1984). This will provide a measure of general performance based on how well the driver maintains a consistent lane position. SDLP has been shown to be among the most important performance measures for evaluating the effects of psychophysiological changes due to impairment from medication use on driving performance (O'Hanlon, 1984).
EEG Measures | Between -0.7 hours and 8 hours post cannabis administration
  Changes in electroencephalogram (EEG) spectral power measures for Delta, Theta, Alpha, Beta, Gamma bands. EEG is sampled at 256 Hertz (Hz) and power spectral measures are calculated in one-second time intervals.
ECG Measures | Between -0.7 hours and 8 hours post cannabis administration
  Changes in heart rate as measured by electrocardiogram (ECG) (R-R interval). ECG is sampled at 256 Hz.

SECONDARY OUTCOMES:
THC Concentration in Plasma Sample | -0.7 hour, 0.25 hour, 1.1 hour, 2 hour, 3 hour, 4.5 hour, 6 hour, 8 hour post cannabis administration
  Measurement of THC concentration levels in plasma over the course of each visit compared to that of the other visits.
THC Concentration Levels in Whole Blood | -0.7 hour, 0.25 hour, 1.1 hour, 2 hour, 3 hour, 4.5 hour, 6 hour, 8 hour post cannabis administration
  Measurement of THC concentration levels in whole blood over the course of each visit compared to that of the other visits.
Event-Related EEG Amplitude | From 0.5 hours to 1.5 hours post cannabis administration
  For each neurocognitive task, EEG will be recorded concurrently. There is a processing pipeline for measuring event-related potentials. This processing pipeline involves pre-processing, artifact removal, and averaging EEG evoked potentials in order to derive amplitude in microvolts.
Event-Related EEG Latency | From 0.5 hours to 1.5 hours post cannabis administration
  For each neurocognitive task, EEG will be recorded concurrently. There is a processing pipeline for measuring event-related potentials. This processing pipeline involves pre-processing, artifact removal, and averaging EEG evoked potentials in order to derive latency in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Berka, B.S, Principal Investigator — Advanced Brain Monitoring
Locations (1):
- University of Iowa. National Advanced Driving Simulator, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified driving and dose data will be made available after analyses are complete.
Supporting Information: Study Protocol, ICF
Time Frame: After analysis of data (May 2021).
Access Criteria: Individual requests to the PI.

REFERENCES:
- [Background] O'Hanlon JF. Driving performance under the influence of drugs: rationale for, and application of, a new test. Br J Clin Pharmacol. 1984;18 Suppl 1(Suppl 1):121S-129S. doi: 10.1111/j.1365-2125.1984.tb02590.x. PMID 6525328